CLINICAL TRIAL: NCT02190864
Title: Patient-Defined Treatment Success and Preferences in Stage IV Lung Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nebraska (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, KM Islam, PhD, Principal Investigator, University of Nebraska
Other Study IDs: 318-13-EP
Record Dates: First submitted 2014-07-02; First posted 2014-07-15 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-11

CONDITIONS: Particularly Rural/Urban Residence; Gender; Age; FACT-TOI Scores; Comorbid Conditions
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Our long-term goal is to integrate non-small cell lung cancer patient treatment preferences into clinical treatment planning.

DETAILED DESCRIPTION:
The following specific aims are proposed:

Aim 1: Determine whether individual patients' preferences, characteristics, and treatment experiences affect the definition of treatment success.

Aim 2: Determine how to best predict real-life patients' treatment choices based on patients' preferences of adverse events.

Aim 3: Determine whether physicians are likely to change their oncologic clinical practice after receiving a detailed communication of their patients' preferences of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide consent
* Greater than or equal to 19 years of age
* Diagnosed with stage IV non-small cell lung cancer (NSCLC)
* Able to understand spoken English
* Eligible to undergo chemotherapy for stage IV NSCLC, to include, but not limited to, those who:

  1. have not yet started chemo
  2. are currently undergoing chemo for stage IV NSCLC
  3. have completed first line stage IV NSCLC chemo or progressed to maintenance for stage IV NSCLC within the last 30 days
  4. elect to have chemo elsewhere -- not at one of the study sites
  5. decline chemo

Exclusion Criteria:

* Age <19 years
* Not willing and/or able to provide consent
* Not able to understand spoken English
* Not eligible to undergo chemotherapy for stage IV NSCLC

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed advanced stage non-small cell lung cancer patients with age > 19 years.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Patient-defined "treatment success" | Baseline
  In advanced stage NSCLC patients does patient-defined "treatment success" differ when both survival and patient preferences of adverse events are accounted for, compared to when success is measured solely by survival? And does it also differ based on individual patient characteristics?
Patients' will to experience adverse events | Baseline
  Will the serious adverse events that an advanced stage NSCLC patient is willing to experience as part of his/her treatment differ after a real-life treatment experience, compared to before treatment?

SECONDARY OUTCOMES:
Summary score derived from patient preferences of adverse events | Up to three months
  In advanced stage NSCLC patients, is a summary score derived from patient preferences of adverse events comparable to a real-life treatment scenario?

OTHER OUTCOMES:
Physicians' will to select a treatment | Two years
  Are physicians treating NSCLC patients more likely to select a treatment that matches patients' drug choices when provided standardized, detailed information on patients' preferences of adverse events compared to when they follow regular clinical practice?

CONTACTS AND LOCATIONS:
Overall Officials: KM Munirul Islam, MD, PhD, Principal Investigator — University of Nebraska
Locations (8):
- United States (8):
  - Moffitt Cancer Center, Tampa, Florida
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Saint Francis Cancer Treatment Center, Grand Island, Nebraska
  - Southeast Nebraska Cancer center, Lincoln, Nebraska
  - Callahan Cancer Center of Great Plains Regional Medical Center, North Platte, Nebraska
  - Nebraska-Western Iowa (NWI) VA Health Care System, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Avera Cancer Institute, Sioux Falls, South Dakota

REFERENCES:
- See also: Patient Centered Outcomes Research Institute — http://pcori.org/
- See also: University of Nebraska Medical Center — http://www.unmc.edu/